Supplementary Analyses for: Comparison of Pro-Inflammatory Cytokines and Bone Metabolism Mediators Around Laser-Lok and Machined Transmucosal Abutments: A Pilot, Randomized Clinical Trial

Prepared for Christopher A. Barwacz, DDS, FAGD (PI) by
Anne Welhaven, MS
Derek R. Blanchette, MS
Xian Jin Xie, PhD
in the Division of Biostatistics and Computational Biology

NCT03572244 8/7/2018

# **Table of Contents**

| Statistical Methods | 3 |
|--------------------------------------------------------|----|
| Comparison of GCF to PICF | 3 |
| Aim 1: Do cytokine levels differ between GCF and PICF? | 4 |
| Descriptive Statistics | 4 |
| Boxplots | 5 |
| GCF and PICF Comparisons | 12 |
| Conclusion for GF and PICF Comparisons | 12 |

#### Statistical Methods

#### Comparison of GCF to PICF

Log-cytokine values were compared between natural teeth and implants using the paired T-test and the Wilcoxon Signed Rank test. Descriptive statistics were prepared to aid interpretation.

P-values were adjusted for multiple comparisons using the Holm (1979)<sup>1</sup> method. All analyses were performed using R 3.4.2 (Vienna, Austria) and SAS 9.4 (Cary, NC) at the 5% level of significance.

<sup>1</sup> Holm, S. (1979). A simple sequentially rejective multiple test procedure. Scandinavian Journal of Statistics, 6, 65–70. http://www.jstor.org/stable/4615733.

# Aim 1: Do cytokine levels differ between GCF and PICF?

# Descriptive Statistics

| Table 1. Descriptive Statistics (PICF – GCF) | | | | | | |
|---|---|---|---|---|---|---|
| Variable | N | Mean | Std Dev | Median | Minimum | Maximum |
| TNFa | 12 | -0.09 | 1.07 | 0.15 | -2.23 | 1.97 |
| IL6 | 12 | -0.38 | 0.74 | -0.21 | -2.50 | 0.35 |
| IL8 | 12 | -0.27 | 1.32 | -0.23 | -2.52 | 1.91 |
| MMP1 | 12 | -0.11 | 0.76 | -0.08 | -1.22 | 1.25 |
| IP10 | 12 | -0.28 | 1.05 | -0.25 | -3.02 | 0.93 |
| MMP8b | 12 | -0.14 | 0.71 | -0.08 | -1.18 | 0.99 |
| IL_1B | 12 | 0.17 | 0.92 | 0.06 | -1.67 | 2.15 |
| MMP13 | 12 | 0.34 | 1.70 | 0.34 | -2.30 | 4.70 |
| ENA78 | 12 | -0.18 | 0.76 | 0.01 | -1.84 | 0.70 |
| MIG | 12 | -0.12 | 0.34 | -0.03 | -0.78 | 0.52 |
| Osteopontin | 12 | -0.22 | 1.24 | 0.04 | -2.47 | 1.76 |
| ITAC1 | 12 | 0.19 | 1.03 | 0.26 | -1.92 | 2.45 |
| Osteoprotegerin | 12 | -0.12 | 1.18 | -0.10 | -2.53 | 2.72 |

# Boxplots



























## GCF and PICF Comparisons

| Table 2. Two-Sample Tests Comparing PICF Cytokine Levels | | | | | |
|---|---|---|---|---|---|
| | | | T-test | Wilcoxon Signed Rank | |
| Measurement | N | P-value | Adjusted P-value | P-value | Adjusted p-value |
| TNFa | 12 | 0.7648 | 0.7648 | 0.9097 | 0.9097 |
| IL6 | 12 | 0.1063 | 0.7199 | 0.0425 | 0.5525 |
| IL8 | 12 | 0.5011 | 0.7199 | 0.5186 | 0.9097 |
| MMP1 | 12 | 0.6428 | 0.7596 | 0.7334 | 0.9097 |
| IP10 | 12 | 0.3760 | 0.7199 | 0.5693 | 0.9097 |
| MMP8b | 12 | 0.4930 | 0.7199 | 0.3804 | 0.9097 |
| IL-1B | 12 | 0.5294 | 0.7199 | 0.6221 | 0.9097 |
| MMP13 | 12 | 0.5060 | 0.7199 | 0.7334 | 0.9097 |
| ENA78 | 12 | 0.4302 | 0.7199 | 0.7910 | 0.9097 |
| MIG | 12 | 0.2323 | 0.7199 | 0.3394 | 0.9097 |
| Osteopontin | 12 | 0.5538 | 0.7199 | 0.8501 | 0.9097 |
| ITAC1 | 12 | 0.5357 | 0.7199 | 0.3911 | 0.9097 |
| Osteoprotegerin | 12 | 0.7268 | 0.7648 | 0.4697 | 0.9097 |

### Conclusion for GF and PICF Comparisons

Before adjustment, the Wilcoxon Signed Rank test found that IL6 was higher in GCF (P = 0.0425).

After adjustment, no significant differences were detected.

Supplementary Analyses for: Comparison of Pro-Inflammatory Cytokines and Bone Metabolism Mediators Around Laser-Lok and Machined Transmucosal Abutments: A Pilot, Randomized Clinical Trial

Prepared for Christopher A. Barwacz, DDS, FAGD (PI) by
Anne Welhaven, MS
Derek R. Blanchette, MS
Xian Jin Xie, PhD
in the Division of Biostatistics and Computational Biology

NCT03572244 7/5/2018

## Contents

| Statistical Methods | 3 |
|---|---|
| Comparison of PICF | 3 |
| Comparison of GCF | 3 |
| Cluster Analyses | 3 |
| Aim 1: Do the cytokine levels of the Laser-Lok PICF differ from the Machined PICF? | 4 |
| Descriptive Statistics | 4 |
| Box Plots | 5 |
| Group Differences | 18 |
| Conclusion for Laser-Lok and Machined PICF Comparisons | 18 |
| Aim 2: Do the cytokine levels of the Laser-Lok GCF differ from the Machined GCF? | 19 |
| Descriptive Statistics | 19 |
| Box Plots | 20 |
| Group Differences | 33 |
| Conclusion for Laser-Lok and Machined GCF Comparisons | 33 |
| Cluster Analysis | 34 |
| Implant Values | 34 |
| Natural Teeth Values | 36 |

#### Statistical Methods

#### Comparison of PICF

Log-cytokine values were compared between the Laser-Lok and Machined implants using the two sample T-test and the Wilcoxon Rank Sum test. Descriptive statistics and box plots were prepared to aid interpretation.

#### Comparison of GCF

Log-cytokine values were compared between the groups of natural teeth using the two sample T-test and the Wilcoxon Rank Sum test. Descriptive statistics and box plots were prepared to aid interpretation.

#### **Cluster Analyses**

Exploratory cluster analyses were performed for subjects and cytokines using the implant values and the natural tooth values (separately). Hierarchical clustering with agglomeration via complete linkage was performed on dissimilarity measures based on Euclidean distances.

P-values were adjusted for multiple comparisons using the Holm (1979)<sup>1</sup> method. All analyses were performed using R 3.4.2 (Vienna, Austria) and SAS 9.4 (Cary, NC) at the 5% level of significance. Analyses were performed using the log-transformed values.

<sup>&</sup>lt;sup>1</sup> Holm, S. (1979). A simple sequentially rejective multiple test procedure. Scandinavian Journal of Statistics, 6, 65–70. http://www.jstor.org/stable/4615733.

# Aim 1: Do the cytokine levels of the Laser-Lok PICF differ from the Machined PICF?

## **Descriptive Statistics**

| Table 1. Descriptive Statistics for PICF Cytokine Levels | | | | | | | |
|---|---|---|---|---|---|---|---|
| Implant | Variable | N | Mean | Std Dev | Median | Minimum | Maximum |
| Laser-Lok | logTNFa | 6 | 2.25 | 1.18 | 2.76 | 0.59 | 3.47 |
| | logIL6 | 6 | 1.80 | 0.31 | 1.84 | 1.38 | 2.12 |
| | logIL8 | 6 | 6.54 | 0.60 | 6.54 | 5.69 | 7.32 |
| | logMMP1 | 6 | 4.48 | 0.64 | 4.37 | 3.76 | 5.51 |
| | logIP10 | 6 | 1.29 | 0.79 | 1.09 | 0.43 | 2.30 |
| | logMMP8b | 6 | 11.37 | 0.37 | 11.38 | 10.77 | 11.90 |
| | logIL_1B | 6 | 5.19 | 0.61 | 5.26 | 4.29 | 5.91 |
| | logMMP13 | 6 | 5.73 | 0.94 | 5.52 | 4.60 | 7.14 |
| | logENA78 | 6 | 4.05 | 0.53 | 3.97 | 3.52 | 4.97 |
| | logMIG | 6 | 6.95 | 0.12 | 6.98 | 6.76 | 7.07 |
| | logOsteopontin | 6 | 6.44 | 1.19 | 6.90 | 4.01 | 7.03 |
| | logITAC1 | 6 | 2.53 | 0.36 | 2.35 | 2.21 | 3.07 |
| | logOsteoprotegerin | 6 | 2.94 | 0.95 | 2.68 | 1.93 | 4.45 |
| Machined | logTNFa | 6 | 2.15 | 1.00 | 1.94 | 1.10 | 3.64 |
| | logIL6 | 6 | 1.61 | 0.36 | 1.71 | 0.94 | 1.92 |
| | logIL8 | 6 | 5.52 | 1.06 | 5.74 | 3.75 | 6.48 |
| | logMMP1 | 6 | 3.89 | 0.72 | 3.98 | 2.58 | 4.69 |
| | logIP10 | 6 | 1.32 | 1.09 | 1.36 | -0.41 | 2.90 |
| | logMMP8b | 6 | 10.61 | 1.11 | 10.58 | 8.84 | 11.88 |
| | logIL_1B | 6 | 4.92 | 1.08 | 4.57 | 3.74 | 6.66 |
| | logMMP13 | 6 | 5.78 | 1.08 | 6.11 | 3.69 | 6.77 |
| | logENA78 | 6 | 3.27 | 0.65 | 3.51 | 1.98 | 3.69 |
| | logMIG | 6 | 6.63 | 0.51 | 6.68 | 5.72 | 7.16 |
| | logOsteopontin | 6 | 6.50 | 0.96 | 6.54 | 5.30 | 7.67 |
| | logITAC1 | 6 | 2.56 | 0.84 | 2.32 | 1.94 | 4.10 |
| | logOsteoprotegerin | 6 | 3.38 | 1.06 | 3.38 | 1.91 | 4.68 |

## **Box Plots**



























# **Group Differences**

| Table 2. Two-Sample Tests Comparing PICF Cytokine Levels | | | | | |
|---|---|---|---|---|---|
| | | Two S | ample T-test | Wilcoxon Rank Sum test | |
| Measurement | N | P-value | Adjusted P-<br>value | P-value | Adjusted p-<br>value |
| TNFa | 12 | 0.8881 | 0.9509 | 0.9376 | 0.9376 |
| IL6 | 12 | 0.3605 | 0.7811 | 0.4862 | 0.8470 |
| IL8 | 12 | 0.0656 | 0.4264 | 0.1208 | 0.7852 |
| MMP1 | 12 | 0.1645 | 0.4277 | 0.2550 | 0.8288 |
| IP10 | 12 | 0.9509 | 0.9509 | 0.9376 | 0.9376 |
| MMP8b | 12 | 0.1425 | 0.4277 | 0.2550 | 0.8288 |
| IL-1B | 12 | 0.6089 | 0.9509 | 0.5864 | 0.8470 |
| MMP13 | 12 | 0.9367 | 0.9509 | 0.8146 | 0.9376 |
| ENA78 | 12 | 0.0456 | 0.4264 | 0.0927 | 0.7852 |
| MIG | 12 | 0.1606 | 0.4277 | 0.3203 | 0.8328 |
| Osteopontin | 12 | 0.9256 | 0.9509 | 0.6966 | 0.9056 |
| ITAC1 | 12 | 0.9232 | 0.9509 | 0.5851 | 0.8470 |
| Osteoprotegerin | 12 | 0.4673 | 0.8678 | 0.4862 | 0.8470 |

### Conclusion for Laser-Lok and Machined PICF Comparisons

There was not enough evidence of a statistically significant difference between Laser-Lok and machined implants for any of the 13 outcomes measured.

# Aim 2: Do the cytokine levels of the Laser-Lok GCF differ from the Machined GCF?

## **Descriptive Statistics**

| Table 3. Descriptive Statistics for GCF Cytokine Levels | | | | | | | |
|---|---|---|---|---|---|---|---|
| Natural Tooth | Variable | N | Mean | Std Dev | Median | Minimum | Maximum |
| Laser-Lok-NT | logTNFa | 6 | 2.52 | 0.50 | 2.47 | 1.80 | 3.28 |
| | logIL6 | 6 | 1.86 | 0.09 | 1.87 | 1.71 | 1.97 |
| | logIL8 | 6 | 6.30 | 0.84 | 5.96 | 5.41 | 7.69 |
| | logMMP1 | 6 | 4.12 | 0.35 | 4.21 | 3.63 | 4.48 |
| | logIP10 | 6 | 1.13 | 0.84 | 0.94 | 0.36 | 2.58 |
| | logMMP8b | 6 | 11.10 | 0.50 | 11.03 | 10.32 | 11.79 |
| | logIL_1B | 6 | 4.70 | 0.82 | 4.91 | 3.24 | 5.51 |
| | logMMP13 | 6 | 5.63 | 0.36 | 5.53 | 5.15 | 6.08 |
| | logENA78 | 6 | 3.94 | 0.79 | 3.61 | 3.52 | 5.53 |
| | logMIG | 6 | 6.88 | 0.18 | 6.93 | 6.55 | 7.03 |
| | logOsteopontin | 6 | 6.82 | 0.49 | 6.88 | 6.28 | 7.60 |
| | logITAC1 | 6 | 2.48 | 0.20 | 2.50 | 2.21 | 2.69 |
| | logOsteoproteger | 6 | 2.84 | 1.56 | 2.84 | 0.51 | 4.86 |
| | in | | | | | | |
| Machined-NT | logTNFa | 6 | 2.13 | 1.15 | 2.10 | 0.59 | 4.04 |
| | logIL6 | 6 | 2.39 | 1.06 | 1.98 | 1.82 | 4.55 |
| | logIL8 | 6 | 6.29 | 1.31 | 5.71 | 5.10 | 8.30 |
| | logMMP1 | 6 | 4.47 | 0.62 | 4.32 | 3.86 | 5.56 |
| | logIP10 | 6 | 2.05 | 2.14 | 1.64 | 0.03 | 5.97 |
| | logMMP8b | 6 | 11.17 | 0.76 | 11.43 | 10.03 | 11.84 |
| | logIL_1B | 6 | 5.06 | 0.80 | 5.05 | 4.00 | 6.02 |
| | logMMP13 | 6 | 5.18 | 1.87 | 5.91 | 1.39 | 6.32 |
| | logENA78 | 6 | 3.75 | 0.68 | 3.62 | 2.98 | 4.75 |
| | logMIG | 6 | 6.95 | 0.32 | 7.06 | 6.49 | 7.31 |
| | logOsteopontin | 6 | 6.56 | 1.21 | 6.81 | 4.23 | 7.78 |
| | logITAC1 | 6 | 2.18 | 1.01 | 2.00 | 1.10 | 3.97 |
| | logOsteoproteger | 6 | 3.69 | 0.82 | 3.94 | 2.42 | 4.42 |
| | in | | | | | | |

## **Box Plots**


























## **Group Differences**

| Table 4. Two-Sample Tests Comparing GCF Cytokine Levels | | | | | |
|---|---|---|---|---|---|
| | | Two Sample T-test | | Wilcoxon Rank Sum test | |
| Measurement | N | P-value | Adjusted P-<br>value | P-value | Adjusted p-<br>value |
| TNFa | 12 | 0.4672 | 0.7783 | 0.3203 | 0.7547 |
| IL6 | 12 | 0.2455 | 0.7783 | 0.0927 | 0.7547 |
| IL8 | 12 | 0.9943 | 0.9943 | 0.4862 | 0.7547 |
| MMP1 | 12 | 0.2584 | 0.7783 | 0.4862 | 0.7547 |
| IP10 | 12 | 0.3485 | 0.7783 | 0.6966 | 0.7547 |
| MMP8b | 12 | 0.8545 | 0.9257 | 0.5864 | 0.7547 |
| IL-1B | 12 | 0.4635 | 0.7783 | 0.4862 | 0.7547 |
| MMP13 | 12 | 0.5739 | 0.7783 | 0.5864 | 0.7547 |
| ENA78 | 12 | 0.6586 | 0.7783 | 0.6966 | 0.7547 |
| MIG | 12 | 0.6387 | 0.7783 | 0.4862 | 0.7547 |
| Osteopontin | 12 | 0.6308 | 0.7783 | 0.9376 | 0.9376 |
| ITAC1 | 12 | 0.5022 | 0.7783 | 0.2007 | 0.7547 |
| Osteoprotegerin | 12 | 0.2660 | 0.7783 | 0.3195 | 0.7547 |

## Conclusion for Laser-Lok and Machined GCF Comparisons

There was not enough evidence of a statistically significant difference between Laser-Lok natural teeth and machined natural teeth for any of the 13 outcomes measured.

# **Cluster Analysis**

### **Implant Values**



Figure 1. Implants: Clustering of subjects based on Euclidean Distance and Log Scaled Values

Clustering of subjects and the resulting dendrogram is given in Figure 1. The tree was partitioned into three clusters and labeled using patient IDs and group assignments.



Figure 2. Implants: Clustering of Cytokines based on Euclidean Distance and Log Scaled Values

Cytokines were clustered and the resulting dendrogram is given in Figure 2. The tree was partitioned into three clusters and labeled using the cytokine names.

#### **Natural Teeth Values**



Figure 3. Natural Teeth: Clustering of subjects based on Euclidean Distance and Log Scaled Values

Clustering of subjects and the resulting dendrogram is given in Figure 1. The tree was partitioned into three clusters and labeled using patient IDs and group assignments.



Figure 4. Natural Teeth: Clustering of Cytokines based on Euclidean Distance and Log Scaled Values

Cytokines were clustered and the resulting dendrogram is given in Figure 2. The tree was partitioned into three clusters and labeled using the cytokine names.